CLINICAL TRIAL: NCT02106793
Title: Comparing Effect of Mitomicin C Versus Placebo for Prevention of Postoperative Endoscopic Sinus Surgery Synechia and Impact on Quality of Life in Thai Patients With Chronic Rhinosinusitis
Brief Title: Mitomicin C for Prevention Postoperative Endoscopic Sinus Surgery Synechia and QOL in Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MitomicinC_PostopESS
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Chronic Rhinosinusitis; Postoperative Nasal Synerchia
Keywords: Chronic Rhinosinusitis; Mitomicin C; Postoperative nasal synerchia
MeSH Terms: interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitomicin C (Experimental): Mitomicin C (0.4 mg/ml) will be provided in a sterile vial and prepared by pharmacist at the Faculty of Medicine Ramathibodi Hospital.The treatment solution will be drawn and soaked ono two one inch neurosurgical cotton pledgets. Each pledget will be placed on each side of the nose for 5 minutes. The nurse will set the alarm for removal of the cotton pledgets, then normal saline will be used to irrigate both sides of the nose, using 100 ml on each side.
  Interventions: Drug: Mitomicin C
- Placebo (Placebo Comparator): Identical placebo solution
  Interventions: Drug: Identical placebo solution

INTERVENTIONS:
Drug: Mitomicin C — Mitomicin C (0.4 mg/ml) will be provided in a sterile vial and prepared by pharmacist at the Faculty of Medicine Ramathibodi Hospital.The treatment solution will be drawn and soaked ono two one inch neurosurgical cotton pledgets. Each pledget will be placed on each side of the nose for 5 minutes. The nurse will set the alarm for removal of the cotton pledgets, then normal saline will be used to irrigate both sides of the nose, using 100 ml on each side.
  Other Names: Mitomycin C
  Arms: Mitomicin C
Drug: Identical placebo solution — Identical placebo solution
  Arms: Placebo

SUMMARY:
Primary objective

* To compare the incidence of postoperative nasal synerchia between Mitomicin C and placebo in patients at 6 months after endoscopic sinus surgery
* To validate the Thai version of disease-specific quality of life tool SNOT-22

Secondary objectives

* To compare the clinical signs and symptoms of CRS in patients who receive Mitomicin C with those who receive placebo
* To compare the disease-specific quality of life in patients who receive Mitomicin C with those who receive placebo
* To compare the side effects of Mitomicin C versus placebo

ELIGIBILITY:
Inclusion Criteria:

* All Thai adults (18 years and older) patients undergoing bilateral endoscopic sinus surgery for CRS
* Patients must not have following diseases or conditions

  * Cystic fibrosis based on positive sweat test or DNA test
  * Gross immunodeficiency (congenital or acquired)
  * Congenital mucociliary problem (eg. Primary ciliary dyskinesia)
  * Altered immune function such as patients with systemic vasculitis, systemic lupus erythematosus, end stage renal disease, cirrhosis, currently taking immunosuppressant or granulomatous disease
  * Severe comorbidity with life expectancy of less than 1 year, such as advanced stage malignancy patient, or severe infection
* Patients are willing to participate and provide written informed consent

Exclusion Criteria:

(None)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Synerchia | 1 year
  The primary outcome of interest is time to event, with the event as the occurrence of nasal synechia. The date of surgery will be used as the beginning date, and the last date will be the date that patient was defined as synechia, or the end of the study period if that patient does not have synechia on follow up.

SECONDARY OUTCOMES:
Scoring of SNOT-22 | 1 year
  Scoring of translated SNOT-22 disease-specific quality of life measurement
Clinical Symptom Score | 6 months
  Clinical symptom score of patients, measured by visual analog score which will be given by research nurse for a patient to fill in at baseline, 1 week, 1, 3, and 6 months.
SNOT-22 | 6 months
  Disease-specific quality of life questionnaire SNOT-22 measurement which will be measured at baseline, 1 week, 1, 3, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pawin Numthavaj, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand